CLINICAL TRIAL: NCT04490668
Title: Association of Human Albumin With Anastomotic Leakage After Gastric Cancer Surgery
Brief Title: Human Albumin and Anastomotic Leakage After Gastric Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BIRENDRA KUMAR SAH, Principal investigator, Ruijin Hospital
Other Study IDs: RJ-GC-Postop-complication 3
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Gastric Cancer; Anastomotic Leak
Keywords: Gastric Cancer; Anastomotic leakage; Human albumin
MeSH Terms: conditions — Stomach Neoplasms; Anastomotic Leak | interventions — Serum Albumin, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Human albumin support: Patients who received intravenous human albumin after gastric cancer surgery
  Interventions: Biological: Human albumin
- No human albumin support: Patients who did not receive intravenous human albumin after gastric cancer surgery
  Interventions: Biological: Human albumin

INTERVENTIONS:
Biological: Human albumin — Patients received intravenous human albumin after gastric cancer surgery. Overall quantity of human albumin were recorded.

SUMMARY:
We investigate whether the intravenously administered human albumin is beneficial to prevent anastomotic leakage after gastric cancer surgery.

DETAILED DESCRIPTION:
Anastomotic leakage after gastric cancer surgery is not very common but it is a very critical postoperative complication. Anastomotic leakage severely compromises the recovery after surgery. It increases the overall burden of patients and hospital resources. Postoperative mortality is higher in patients with anastomotic leakage.

Human albumin is routinely administered after surgery with a unproven hypothesis that the human albumin is beneficial to prevent anastomotic leakage. We investigate whether the intravenously administered human albumin is beneficial to prevent anastomotic leakage after gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric cancer
* Patients who underwent radical gastrectomy

Exclusion Criteria:

* Patient who did not undergo gastrectomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastric cancer who underwent gastrectomy with adequate lymph node dissection.
Sampling Method: Non-Probability Sample
Enrollment: 1049 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the rate of anastomotic leakage | Up to one months after the discharge of last patient
  The rate of anastomotic leakage were compared among both groups

CONTACTS AND LOCATIONS:
Overall Officials: Birendra K Sah, PH D, Principal Investigator — Ruijin Hospital; Chen Li, PH D, Study Director — Ruijin Hospital; Zhenggang Zhu, PH D, Study Chair — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No